CLINICAL TRIAL: NCT06922682
Title: The Effect of Providing Pregnant Women Training on Sudden Infant Death Syndrome (SIDS) on the Post-Partum Risky Behaviors: Randomized Controlled Trial
Brief Title: Training About Sudden Infant Death Syndrome
Acronym: Training about
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Hatice Uzşen, Research Assistant, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023/124
Record Dates: First submitted 2025-04-03; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Sudden Infant Death
Keywords: Sudden Infant Death; newborn; mother; risk factors
MeSH Terms: conditions — Sudden Infant Death

STUDY DESIGN:
Intervention Model Description: a parallel group, randomized, controlled experimental study.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Pregnant women in their 38th week of pregnancy and later, who visited the hospital to have their NST scans, were then invited to the training with the Risk Factors Triggering Sudden Infant Death Syndrome Training Booklet
  Interventions: Behavioral: Training with Sudden Infant Death Syndrome Training Booklet
- Control Group (No Intervention): Pregnant women in this group were not provided a specific training on the risk factors triggering sudden infant death syndrome. The clinic has already offered a pregnancy school where routine prenatal care training is provided.

INTERVENTIONS:
Behavioral: Training with Sudden Infant Death Syndrome Training Booklet — Sudden Infant Death Syndrome Training Booklet was prepared. Prgenant women who agreed to participate were provided a face-to-face training on the risk factors triggering sudden infant death syndrome through the booklet. Following the educational session, they received the safe sleep handout to use at home and were informed that the researcher would call them two months later to check on their adherence to safe sleep practices. Following the training, participants were re-administered the Knowledge Level on Sudden Infant Death Syndrome and Risky Behavior Identification Questionnaire and the training booklet was given to them as a gift. Two months after the training, the pregnant women were contacted via phone and they were required to fill out the Knowledge Level on Sudden Infant Death Syndrome and Risky Behavior Identification Questionnaire once again.
  Arms: Intervention Group

SUMMARY:
Sudden infant death syndrome, which constitutes a significant proportion of all infant deaths, is associated with various preventable risk factors. The study aims examine effects of training provided to pregnant women about risk factors triggering sudden infant death syndrome before birth on the post-partum knowledge level and behaviors of mothers.

DETAILED DESCRIPTION:
Sudden infant death syndrome, which constitutes a significant proportion of all infant deaths, is associated with various preventable risk factors. To examine effects of training provided to pregnant women about risk factors triggering sudden infant death syndrome before birth on the post-partum knowledge level and behaviors of mothers. Pre-test post-test designed, randomized controlled, experimental study was conducted in Turkey, 2024. Sixty pregnant women were employed in intervention and control groups. Face-to-face training on risk factors triggering sudden infant death syndrome was provided to pregnant women in intervention group. Study data were collected using "Personal Information Form, Knowledge Level on Sudden Infant Death Syndrome and Risky Behavior Identification Questionnaire". Data were collected face to face before training and after training and via telephone 2 months after training.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who were in the 38th week of their pregnancy and older,
* Lived a healthy pregnancy,
* Had no communication problems,
* Can speak and understand Turkish,
* Agreed to participate in the study were included.

Exclusion Criteria:

* Pregnant women who were earlier than 38 weeks pregnant,
* Had difficulty in communicating,
* Were illiterate and unable to speak Turkish,
* Who filled out the forms incompletely were not included.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Knowledge Level on Sudden Infant Death Syndrome and Risky Behavior Identification Questionnaire | 20 minutes before training, just after training and 2 month later
  Questionnaire, developed by authors consists of 2 sections. First section aims to determine knowledge level of pregnant women about sudden infant death syndrome. Questionnaire consisting of 17 questions are answered as true, false, or I do not know. Items answered as "True" are scored 1 point, whereas items answered as "False" or "I don't know" are scored as 0. Questionnaire includes reverse coded items. The lowest possible score in the questionnaire is 0 and the highest possible score is 17. The second section consists of questions aiming to determine the risky behaviors of pregnant women that may cause sudden infant death syndrome. A total of 26 questions in this section are answered as never (1 point), rarely (2 points), sometimes (3 points), often (4 points) and always (5 points). The questionnaire includes reverse coded items; the lowest and the highest possible scores in the questionnaire are 26 and 130, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Uzsen, PHD, Principal Investigator — Ondokuz Mayis Univeristy
Locations (1):
- Samsun Gynecology and Children's Diseases Hospital in Turkey, Samsun, Black Sea Zone, Turkey (Türkiye)